CLINICAL TRIAL: NCT03264482
Title: Treatment of Benign Prostatic Hyperplasia: High Power Thulium Laser Front Fire Vaporization VS Transurethral Resection - A Randomized Controlled Trial
Brief Title: High Power Thulium Vaporization vs Transurethral Resection of the Prostate for Treatment of BPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Elshal, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THUVAP VS M-TURP
Record Dates: First submitted 2017-08-14; First posted 2017-08-29 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THUVAP (Active Comparator): thulium vaporization
  Interventions: Procedure: THUVAP
- M-TURP (Active Comparator): monopolar transurethral resection
  Interventions: Procedure: M-TURP

INTERVENTIONS:
Procedure: M-TURP — endoscopic resection of the prostatic adenoma
  Arms: M-TURP
Procedure: THUVAP — vaporization of prostatic adenoma via THULIUM laser
  Arms: THUVAP

SUMMARY:
the investigators plan to test Thulium laser vaporization using high power ( 200w ) Front fire vaporization compared to standard M-TURP in reduction of LUTS secondary to BPH in a prospective randomized trial.

DETAILED DESCRIPTION:
When Lower Urinary Tract Symptoms (LUTS) are refractory to medical therapy and bothersome enough to warrant surgical intervention, transurethral resection of the prostate (TURP) has been the historical reference-standard procedures for prostate size between 30-80 ml for years.

Over the past decade, New minimally invasive surgical therapies (MIST), new medications, and novel combinations of medical therapies have expanded the number of treatment options ranging from watchful waiting to open surgery. The range of treatment options is as broad as the BPH spectrum of symptoms.

These treatment options include prostate vaporization, resection and enucleation using various energy sources , however the main theme for all these new procedures that they were done using physiological saline as an irrigant nullifying the risk of TUR syndrome.

One of the biggest changes in surgical treatment of BPH over the past 2 decades has been the introduction and use of lasers. Two-micron (Thulium) continuous-wave (CW) laser may have several advantages, including sufficient homeostasis with minimal thermal injury, more precise tissue incision, and operation in CW/pulsed modes. Pieces of the prostate are vaporized small enough to evacuate through the resectoscope sheath and use of a mechanical tissue morcellator is not required.

The introduction of the latest generation of the Thulium laser namely "200w laser " raises the expectations of the prostate vaporization.

ELIGIBILITY:
Inclusion Criteria:

* Patients' age ≥50 years
* LUTS secondary to BOO due to BPH who failed medical treatment
* International prostate symptom scores (IPSS) >15 and bother score (QOL) ≥ 3 (according to IPSS question 8)
* Peak urinary flow rate (Qmax) <15 ml/sec with at least 125 ml voided volume or Patients with acute urine retention secondary to BPH who failed trial of voiding on medical treatment.
* ASA (American society of anaesthesiologists) score ≤3.
* TRUS prostate size between 30-80 ml

Exclusion Criteria:

* Patient with neurological disorder which might affect bladder function as cerebrovascular stroke, Parkinson disease
* Active urinary tract infection,
* Presence of active bladder pathology (within the last 2 years)
* Known prostate cancer patients will be excluded preoperatively on the basis of digital rectal examination, prostate specific antigen level, and TRUS imaging followed by prostate biopsies if necessary.
* Patient has a disorder of the coagulation cascade (e.g., liver cell failure) or disorders that affect platelet count or function (e.g., von Willebrand disease) that would put the subject at risk for intraoperative or postoperative bleeding.
* Patient is unable to discontinue anticoagulant and antiplatelet therapy preoperatively (3-5 d) except for low-dose aspirin (e.g., 100 mg).
* Patient has had an acute myocardial infarction or open-heart surgery <180 days prior to the date of informed consent

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2018-12-02 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
IPSS score at 12 months . | 12 months
  international prostate symptom score (both voiding & storage symptom subscores )

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M. Elshal, MD, Principal Investigator — Mansoura University
Locations (1):
- Urology and nephrology center, Al Manşūrah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided